CLINICAL TRIAL: NCT05236348
Title: Single-center Prospective Clinical Trial to Validate the Performance of the Aktiia Optical Blood Pressure Monitoring (OBPM) Device at the Wrist Against Double Auscultation
Brief Title: Performance of the Aktiia Optical Blood Pressure Monitoring Device Against Double Auscultation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aktiia SA (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: OBPM_Auscultatory2022
Record Dates: First submitted 2021-12-28; First posted 2022-02-11 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: Hypertension; Blood Pressure; Heart Rate
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Intervention Model Description: All study participants will wear the Aktiia.bracelet-us during 9 visits that will be held over the span of seven days. In order to induce blood pressure changes and to simulate ambulatory scenarios, the study participants will be asked to perform a set of activities, involving body position changes and physical exercises during these visits.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients 21-60yo with Aktiia.product-us (Experimental): All study participants will wear the Aktiia.product-us during 9 visits that will be held over the span of seven days.
  Interventions: Device: Aktiia.product-us
- Patients 60-85yo with Aktiia.product-us (Experimental): All study participants will wear the Aktiia.product-us during 9 visits that will be held over the span of seven days.
  Interventions: Device: Aktiia.product-us

INTERVENTIONS:
Device: Aktiia.product-us — The study will collect data from subjects by means of the device under test and collect data from subjects by means of double-auscultation, pulse oximetry and volume-clamp BP reading while subjects wear the devices at different body positions and induce BP changes, during eight visits that will be held over the span of seven days, and generate performance reports.
  Other Names: Aktiia bracelet; Aktiia product; Aktiia.product

SUMMARY:
This study with N = 225 participants (1 cohort of a minimum of 85 and maximum of 140 participants, and an additional cohort with 85 participants) over 9 visits has been designed to assess the accuracy of Aktiia.product-us systolic and diastolic blood pressure measurements against double-auscultation reference measurements. In order to induce blood pressure changes and to simulate ambulatory scenarios, the study participants will be asked to perform a set of activities, involving body position changes and physical exercises. Additionally, this study will compare the heart rate measured by Aktiia.product-us against the reference readings provided by a finger pulse oximeter (as per ISO80601-2-61). The reliability of the auscultation readings will be controlled with simultaneous volume-clamp measurements.

DETAILED DESCRIPTION:
According to the World Health Organization, by 2025 hypertension will affect 1.5 billion adults worldwide. Half of the adult population suffering from hypertension is currently not diagnosed and half of the treated population is not at the defined target of BP.

Widespread use of out-of-office Blood Pressure measurement is one of the proposed strategies to fight against hypertension worldwide.

Aktiia S.A. has developed an intermittent automated non-invasive cuffless blood pressure monitor, determining the values of the systolic blood pressure, the diastolic blood pressure and the heart rate. This miniature device is comfortably positioned with a bracelet on a user's wrist.

The goal of this study is to establish a reasonable assurance of safety and effectiveness with Aktiia OBPM system for monitoring blood pressure in home use.

In particular, the study will collect data from subjects by means of the device under test and collect data from subjects by means of double-auscultation, pulse oximetry and volume-clamp BP reading while subjects wear the devices at different body positions and induce Blood Pressure changes, during eight visits that will be held over the span of seven days, and generate performance reports.

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects (aged between 21 and 85 years old)
* Subjects can read and speak French
* Subjects can perform simple physical exercises
* Subjects agreeing to attend the totality of 9 visits
* Subjects that have signed the informed consent form

Exclusion Criteria:

* Clinical staff collaborating with study PI
* Subjects with tachycardia (heart rate at rest > 120bpm)
* Subjects with atrial fibrillation
* Subjects with diabetes
* Subjects with renal dysfunctions
* Subjects with hyper-/hypothyroidism
* Subjects with pheochromocytoma
* Subjects with Raynaud's disease
* Subjects with trembling and shivering
* Subjects with interarm systolic difference > 15 mmHg
* Subjects with interarm diastolic difference > 10 mmHg
* Subjects with arm paralysis
* Women in known pregnancy (for ARM 1 only)
* Subjects with an arteriovenous fistula
* Subjects with arm amputations
* Subjects with the upper arm circumference < 22cm or > 42 cm
* Subjects with the wrist circumference > 21 cm
* Subjects with the exfoliative skin diseases
* Subjects with lymphoedema

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 225 (Estimated)
Dates: Start 2022-01-11 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Blood pressure mean value of differences | 1 week
  The mean value of the differences between Aktiia.product-us and double auscultation blood pressure measurements.
Blood pressure standard deviation of differences | 1 week
  The standard deviation of the differences between Aktiia.product-us and double auscultation blood pressure measurements.

SECONDARY OUTCOMES:
Heart rate root-mean-square error | 1 week
  The root-mean-square difference between the Aktiia.product-us heart rate determinations and the reference method.

CONTACTS AND LOCATIONS:
Overall Officials: Gregoire Wuerzner, MD, Principal Investigator — Service of Nephrology and Hypertension CHUV
Locations (1):
- University of Lausanne Hospitals, Lausanne, Switzerland

IPD SHARING:
Plan to Share IPD: No